CLINICAL TRIAL: NCT02396784
Title: A Randomised Controlled Trial for Overweight and Obese Parents to Prevent Childhood Obesity - China
Brief Title: Early Stockholm Obesity Prevention Program (EarlySTOPP-China)
Acronym: EarlySTOPP-CN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jianduan Zhang, Associate professor, Huazhong University of Science and Technology
Other Study IDs: EarlySTOPP-CN
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Overweight; Obesity
Keywords: child overweight; child obesity; prevention; targeted intervention; development of overweight
MeSH Terms: conditions — Overweight; Obesity; Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High risk: One parent has a BMI of greater than or equal to 28, or both parents have a BMI of greater than or equal to 24
- Normal risk: Both parents have a BMI of smaller than 24

SUMMARY:
Early STOPP project promotes good health in children from early age by supporting good habits for the whole family. Our aim is to see if we can prevent overweight and obesity in children in families where parents are overweight or obese. Normal weight parents will also be needed in this study.

Background: Several daily habits lead to less favorable health factors. For example, using the car instead of cycling or walking - leads to less activity in everyday life. Individuals also eat more unhealthy foods in larger portions. In combination with genetics, social in heritage and surrounding factors this contributes to increase overweight and obesity among children not only in adults but also in children.

Good treatment for childhood obesity are lacking, making prevention very important. The earlier good habits are introduced to a child the better it is.

In Early STOPP project we study food, physical activity and sleep habits in the families with a child of one year of age. The height, weight, waist circumference and blood pressure will be recorded in both child and parents. The parents will answer questionnaires about food, physical activity and sleeping habits for both the child and themselves. During the study, the child's physical activity will be measured. Based on our observations we aim to develop the preventive strategies for the families with very young children.

ELIGIBILITY:
Inclusion Criteria:

* one obese or two overweight parents, 1 year old child

Exclusion Criteria:

* weight effecting diseases

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 1-6 yrs
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index score(BMI sds) at the age 6 years | 5 years
  Weight gain, reflected in BMI sds will reflect the difference between two groups (case group and control group)

SECONDARY OUTCOMES:
sleeping hehavior | 5 years
  sleeping duration will be monitored to study its effect
biomarkers | 5 years
  such as bacterial population in feces and in saliva
physical activity and sedentary behavious | 5 years
  physical activity and sedentary behavious will be monitored
dietary intake | 5 years
  changes in dietary habits and behaviour will be monitored
socioeconomic factors | 5 years
  factors effecting obesity development will be assessed in order to understand their impacts

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Sobko, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Tongji Medical College, Wuhan, Hubei, China